CLINICAL TRIAL: NCT06294275
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, and Pharmacokinetics of LP-001 Injection in Healthy Subjects Following Single and Multiple Doses
Brief Title: A Study of Single and Multiple Dose Administration of LP-001 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Longbio Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P-10-LP001-2022-01
Record Dates: First submitted 2024-02-20; First posted 2024-03-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Single Person

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cohort 1: LP-001 Dose 1 (Single) (Experimental): Single dose administration of LP-001 with dose 1
  Interventions: Biological: LP-001 Dose 1 (Single)
- Cohort 2: LP-001 Dose 2 (Single) (Experimental): Single dose administration of LP-001 with dose 2
  Interventions: Biological: LP-001 Dose 2 (Single)
- Cohort 3: LP-001 Dose 3 (Single) (Experimental): Single dose administration of LP-001 with dose 3
  Interventions: Biological: LP-001 Dose 3 (Single)
- Cohort 4: LP-001 Dose 4 (Single) (Experimental): Single dose administration of LP-001 with dose 4
  Interventions: Biological: LP-001 Dose 4 (Single)
- Cohort 5: LP-001 Dose 5 (Single) (Experimental): Single dose administration of LP-001 with dose 5
  Interventions: Biological: LP-001 Dose 5 (Single)
- Cohort 6: LP-001 Dose 6 (Single) (Experimental): Single dose administration of LP-001 with dose 6
  Interventions: Biological: LP-001 Dose 6 (Single)
- Cohort 7: Placebo (Single) (Placebo Comparator): Single dose administration of placebo drug
  Interventions: Biological: Placebo (Single)
- Cohort 8: LP-001 Dose 7 (Multiple) (Experimental): LP-001 with dose 7 was administered 4 times in total
  Interventions: Biological: LP-001 Dose 7 (Multiple)
- Cohort 9: LP-001 Dose 8 (Multiple) (Experimental): LP-001 with dose 8 was administered 4 times in total
  Interventions: Biological: LP-001 Dose 8 (Multiple)
- Cohort 10: Placebo (Multiple) (Placebo Comparator): Placebo drug was administered 4 times in total
  Interventions: Biological: Placebo (Multiple)

INTERVENTIONS:
Biological: LP-001 Dose 1 (Single) — A single dose of LP-001 (Dose 1) was administered subcutaneously.
  Arms: Cohort 1: LP-001 Dose 1 (Single)
Biological: LP-001 Dose 2 (Single) — A single dose of LP-001 (Dose 2) was administered subcutaneously.
  Arms: Cohort 2: LP-001 Dose 2 (Single)
Biological: LP-001 Dose 3 (Single) — A single dose of LP-001 (Dose 3) was administered subcutaneously.
  Arms: Cohort 3: LP-001 Dose 3 (Single)
Biological: LP-001 Dose 4 (Single) — A single dose of LP-001 (Dose 4) was administered subcutaneously.
  Arms: Cohort 4: LP-001 Dose 4 (Single)
Biological: LP-001 Dose 5 (Single) — A single dose of LP-001 (Dose 5) was administered subcutaneously.
  Arms: Cohort 5: LP-001 Dose 5 (Single)
Biological: LP-001 Dose 6 (Single) — A single dose of LP-001 (Dose 6) was administered subcutaneously.
  Arms: Cohort 6: LP-001 Dose 6 (Single)
Biological: Placebo (Single) — A single dose of placebo was administered subcutaneously.
  Arms: Cohort 7: Placebo (Single)
Biological: LP-001 Dose 7 (Multiple) — LP-001 (Dose 7) was administered multiple times subcutaneously.
  Arms: Cohort 8: LP-001 Dose 7 (Multiple)
Biological: LP-001 Dose 8 (Multiple) — LP-001 (Dose 8) was administered multiple times subcutaneously.
  Arms: Cohort 9: LP-001 Dose 8 (Multiple)
Biological: Placebo (Multiple) — Placebo was administered multiple times subcutaneously.
  Arms: Cohort 10: Placebo (Multiple)

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, immunogenicity, pharmacokinetics, pharmacodynamics, and efficacy of LP-001 in healthy volunteers. The study will be conducted in 2 parts: Part 1, the single ascending dose (SAD) is the first in human (FIH) study of LP-001 and Part 2, multiple ascending dose (MAD).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females aged 18 through 50 years.
2. Male subjects with a weight of ≥50 kg, female subjects with a weight of ≥45 kg, and BMI between 19.0 and 26.0 kg/m² (inclusive).
3. Male subjects and their partners, or female subjects, must agree to use one or more non-pharmacological contraceptive measures during the trial and up to 6 months after the end of the trial (such as complete abstinence, condoms, intrauterine devices, partner sterilization, etc.), and should have no plans for sperm or egg donation.
4. The upper limits for hemoglobin (Hb) and hematocrit (HCT) are 165 g/L and 49%, respectively, for males, and 150 g/L and 45%, respectively, for females.
5. Subjects have a full understanding of the trial's purpose, nature, methods, and potential adverse reactions, voluntarily agree to participate in the trial, and sign the informed consent form.
6. Subjects can communicate effectively with the researchers and can comply with the study protocol as specified.

Exclusion Criteria:

1. Family history of early-onset coronary artery disease, including first- or second-degree relatives diagnosed with coronary heart disease or angina before the age of 50; any family history of hematological disorders, such as thrombosis or increased clotting risk, or any family history of deep vein thrombosis, pulmonary embolism, stroke, hemolytic anemia, or hemoglobinopathies; family history of hypertension. Alternatively, the subject has a personal medical history of the aforementioned conditions.
2. Presence of liver or kidney diseases or conditions affecting drug absorption, distribution, metabolism, or excretion, including other medical situations such as surgical procedures, trauma, etc. that may interfere with these processes.
3. Diagnosed with malignant tumors or having a history of malignant tumors, excluding non-melanoma skin cancer cured for more than 3 years.
4. HIV testing positive (HIV-Ab), hepatitis B virus (HBV) testing positive (HBsAg or HBcAb), hepatitis C virus (HCV) positive (HCV-RNA), and specific antibodies for syphilis positive, excluding positive results caused by immunization.
5. Abnormal vital signs (reference normal range: sitting systolic blood pressure 90-139 mmHg, diastolic blood pressure 60-89 mmHg, pulse rate 60-100 beats/min; body temperature 35.4-37.7°C) or abnormal electrocardiogram (QTcB≥450 ms), or clinically significant abnormalities in physical examination, laboratory tests, and abdominal ultrasound (as judged by the clinical research doctor).
6. Clear history of drug allergy or specific hypersensitivity reactions (asthma, urticaria, allergic rhinitis, eczematous dermatitis); known allergies to the investigational drug and excipients, or allergies to similar drugs; individuals intolerant to subcutaneous injections or with a history of fainting during needle procedures.
7. Use of erythropoiesis-stimulating agents or treatment with other biologics within the six months prior to screening.
8. Participation in any other drug clinical trial within the 3 months prior to screening or within 5 half-lives of any investigational drug from other clinical trials (selecting the longer time period).
9. Pregnant or lactating women or women with the possibility of becoming pregnant.
10. Any condition deemed unsuitable for participation in the study by the investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-09-03 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Adverse events | Observation for 36 days after administration
  Number of subjects with treatment-related Treatment Emergent Adverse Events (TEAEs).

SECONDARY OUTCOMES:
Time to peak concentration (Tmax) of LP-001 | Observation for 36 days after administration
  The time when the blood drug concentration reaches its peak after a single dose of medication.
Maximum concentration (Cmax) of LP-001 | Observation for 36 days after administration
  The maximum concentration of LP-001 in the bloodstream after administration.
Elimination half-life (t1/2) of LP-001 | Observation for 36 days after administration
  The time required for the concentration of LP-005 in the bloodstream to decrease by half.
Area under the concentration-time curve (AUC0-t) of LP-001 | Observation for 36 days after administration
  The time required for the concentration of LP-005 in the bloodstream to decrease by half.
Apparent clearance rate (CL/F) of LP-001 | Observation for 36 days after administration
  The ratio of drug clearance to drug concentration, represents the apparent clearance of a drug after administration, adjusted for bioavailability.
Assessment of immunogenicity | Observation for 36 days after administration
  The proportion of anti drug antibody (ADA) positive subjects at different detection time points.
Assessment of hemoglobin (Hb) change | Observation for 36 days after administration
  Concentration of Hemoglobin changes from baseline at various time points of assessment.
Assessment of red blood cell (RBC) count change | Observation for 36 days after administration
  The count of RBC changes from baseline at various time points of assessment.
Assessment of reticulocyte (Rtc) count change | Observation for 36 days after administration
  The count of Rtc changes from baseline at various time points of assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, China